CLINICAL TRIAL: NCT00255515
Title: An Open, Randomised, Parallel, Three Treatment Groups, Multicentre, Phase IV Study - in Real Life - to Compare the Change in Social Outcome of Quetiapine Fumarate (Seroquel®) Combined With Cognitive Remediation Therapy to Conventional Treatment in Patients With Schizophrenia.
Brief Title: Seroquel® Combined With Cognitive Remediation Therapy to Conventional Treatment in Patients With Schizophrenia
Acronym: SCORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Birgit Ekholm, MD, Neuroscience, AstraZeneca Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1449L00004; SCORE
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

ARMS (3):
- 1 (Experimental): quetiapine fumarate
  Interventions: Drug: Quetiapine fumarate
- 2 (Active Comparator): Conventional treatment for schizophrenia
  Interventions: Drug: conventional treatment for schizophrenia
- 3 (Experimental): quetiapine fumarate + Cognitive Remediation Therapy
  Interventions: Drug: Quetiapine fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate — oral
  Other Names: Seroquel
  Arms: 1; 3
Drug: conventional treatment for schizophrenia — various standard therapies
  Arms: 2

SUMMARY:
The purpose of this study is to compare efficacy of quetiapine fumarate combined with Cognitive Remediation Therapy (CRT) to conventional treatment by evaluating change in social outcome in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Documented clinical diagnosis of schizophrenia or schizoaffective disorder for at least 2 years.
* Clinically stable and in an outpatient setting before entering the study (visit 1).

Exclusion Criteria:

* Use of clozapine and quetiapine within two months prior to visit 1.
* If total points are ≤ 55 Intelligence quotient (IQ) according to score of WAIS-III test at visit 1.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Social outcome measured by Strauss-Carpenter scale | change from baseline to last visit and end of CRT

SECONDARY OUTCOMES:
Change in PANSS total score | change from baseline to visit 2, from baseline to end of CRT and from baseline to last visit
Change in PANSS positive, negative and general psychopathology symptom subscales | change from baseline to visit 2, from baseline to end of CRT and from baseline to last visit
Change in cognition as measured by a Cognitive Battery of Tests | change from baseline to end of CRT and from baseline to last visit

CONTACTS AND LOCATIONS:
Overall Officials: Leif Lindström,, Principal Investigator — Västerås
Locations (15):
- Sweden (15):
  - Research Site, Eskilstuna
  - Research Site, Gothenburg
  - Research Site, Hisingsbacka
  - Research Site, Huddinge
  - Research Site, Jönköping
  - Research Site, Lidingö
  - Research Site, Limhamn
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Norsborg
  - Research Site, Nyköping
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Umeå
  - Research Site, Västerås